CLINICAL TRIAL: NCT03340623
Title: Use of the Venous Coupler in Breast Reconstruction by Means of a Deep Inferior Epigastric Perforator: Reduction of Surgery Length and Venous Thromboses ?
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Socorro ORTIZ, Head of clinic, Brugmann University Hospital
Other Study IDs: CHUB-venous coupler
Record Dates: First submitted 2017-11-09; First posted 2017-11-13 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Mammary Reconstruction
Keywords: DIEP; Venous coupler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mammary reconstruction by DIEP with venous coupler
  Interventions: Device: Venous coupler
- Mammary reconstruction by DIEP without venous coupler

INTERVENTIONS:
Device: Venous coupler — A coupler can be used to perform a venous anastomosis. It is a double ring with pins on only one of its 2 faces. The technique consists in clamping the two veins, estimating the intima-to-intimal diameter of the vessels, choosing the coupler of the appropriate size, sliding the vein in the ring and evers the edges of the vessel to fix them on the pins, redo the same thing for the other vein and finally bring the two vessels together in order to clip them together.
  Groups: Mammary reconstruction by DIEP with venous coupler

SUMMARY:
This is a retrospective study performed on medical records, in order to compare the number of venous thromboses, the surgery duration, the complications rate and the duration of anastomosis in breast reconstructive surgeries by the DIEP (Deep Inferior Epigastric Perforator Flap) technique, with or without the use of a venous coupler.

DETAILED DESCRIPTION:
Breast cancer is the most common and deadliest cancer among women in Belgium. Women with invasive cancer may be offered a total mastectomy with or without adjuvant/neoadjuvant therapy, and with or without breast reconstruction. It is obvious that the loss of a breast can impact the self-image, hence the importance of informing the patient about the possibilities of breast reconstruction. Between 14 and 20% of women choose to resort to reconstruction.

Different types of breast reconstruction exist: prosthetic reconstruction, lipolifting and flap reconstruction (of large dorsal, gluteus maximus, rectus abdominis muscle and "DIEP").

DIEP (Deep Inferior Epigastric Perforator Flap) presents numerous advantages. It consists in the use of a free cutaneo-greasy flap taken from the abdomen, without muscle removed. The abdominal skin has a similar appearance to the breast skin and, thanks to the presence of fat, the missing volume is replaced by a living tissue. Weakness of the abdominal wall is also avoided. However, it remains a surgical procedure with possible complications.

There are several steps in this surgery. The first is to dissect the abdominal flap by talking the skin and subcutaneous fat and isolating one or two branches of the lower epigastric artery and one or two veins. The donor area is then closed. The second step is to prepare the recipient area, ie dissect the artery that will be anastomosed with the lower deep epigastric artery.This artery can be the intern mammary artery, the thoraco-dorsal artery or more rarely the axillary artery. The third step consists of performing arterial and venous anastomoses and checking the quality of these.

Two microanastomoses must thus be performed: arterial and venous. The classic technique, the most used, is to suture the 2 veins. Alternatively, a coupler device can be used to perform the venous anastomosis.

It is therefore interesting to compare the classical method and the venous coupler method in terms of surgery duration, venous thrombosis and complications. If the coupler is proved effective, it could replace the manual suture.

Venous thrombosis is the main cause of flap failure. But surgery duration has also an impact on the complication rate, and the anastomosis duration corresponds to the time during which the flap is not perfused. It is thus necessary to keep it to a minimum in order to reduce the risk of flap loss.

ELIGIBILITY:
Inclusion Criteria:

* Total mastectomy with mammary reconstruction by the DIEP technique
* Patients treated within the CHU Brugmann Hospital
* Patients treated between 01/01/2017 and 01/09/2017

Exclusion Criteria:

/

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women having had a total mastectomy and a mammary reconstruction by the DIEP technique with or without venous coupler utilisation, treated within the CHU Brugmann hospital between 01/01/2017 and 01/09/2017.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Rate of venous thrombosis | Up to 1 week after mammary reconstruction surgery
  Rate of venous thrombosis
Surgery duration | At the date of mammary reconstruction surgery.
  Duration of the mammary reconstruction surgery with the DIEP technique
Anastomosis duration | At the date of mammary reconstruction surgery.
  Duration of the anastomosis during the mammary reconstruction surgery

SECONDARY OUTCOMES:
Age | At the date of mammary reconstruction surgery.
  Patient age
Body mass index | At the date of mammary reconstruction surgery.
  Body mass index
Tabagism | At the date of mammary reconstruction surgery.
  Tabagism status (smoker/non smoker)
Co-morbidity : diabetes | At the date of mammary reconstruction surgery.
  Medical history of diabetes
Co-morbidity : cardio-vascular disease | At the date of mammary reconstruction surgery.
  Medical history of cardio-vascular disease
Co-morbidity : medical history of venous thrombosis | At the date of mammary reconstruction surgery.
  Medical history of venous thrombosis
Immediate of differed reconstruction | At the date of mammary reconstruction surgery.
  Reconstruction performed immediately after mastectomy or not
Unilateral or Bilateral DIEP | At the date of mammary reconstruction surgery.
  Unilateral or Bilateral DIEP
Medical complications (yes/no) | Up to one week after mammary reconstruction surgery
  Medical complications within the grafted flap
Type of cancer treatment | At the date of mammary reconstruction surgery.
  (neo)adjuvant chemiotherapy or (neo)adjuvant radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Miszewska, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Camara O, Herrmann J, Egbe A, Koch I, Gajda M, Runnebaum IB. Venous coupler for free-flap anastomosis. Anticancer Res. 2009 Jul;29(7):2827-30. PMID 19596969
- [Background] Kulkarni AR, Mehrara BJ, Pusic AL, Cordeiro PG, Matros E, McCarthy CM, Disa JJ. Venous Thrombosis in Handsewn versus Coupled Venous Anastomoses in 857 Consecutive Breast Free Flaps. J Reconstr Microsurg. 2016 Mar;32(3):178-82. doi: 10.1055/s-0035-1563737. Epub 2015 Sep 15. PMID 26372685
- [Background] Rozen WM, Whitaker IS, Acosta R. Venous coupler for free-flap anastomosis: outcomes of 1,000 cases. Anticancer Res. 2010 Apr;30(4):1293-4. PMID 20530442
- See also: Related Info — http://www.think-pink.be/